CLINICAL TRIAL: NCT02016911
Title: Investigation of Pharmacokinetics, Safety and Tolerability of Oral Semaglutide (NNC0113-0217) in Subjects With Mild, Moderate and Severe Degrees of Hepatic Impairment Compared to Subjects With Normal Hepatic Function
Brief Title: Pharmacokinetics, Safety and Tolerability of Oral Semaglutide in Subjects With Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9924-4082; 2013-000550-21 (EudraCT Number); U1111-1139-1272 (Other: WHO)
Record Dates: First submitted 2013-12-12; First posted 2013-12-20 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2; Healthy
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subjects with hepatic impairment (Experimental)
  Interventions: Drug: semaglutide
- Subjects with normal hepatic function (Active Comparator)
  Interventions: Drug: semaglutide

INTERVENTIONS:
Drug: semaglutide — Once daily oral administration of semaglutide formulated with SNAC. Dose escalation, with 5 days on 5 mg followed by 5 days on 10 mg

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to investigate the pharmacokinetics (the exposure of the trial drug in the body), safety and tolerability of oral semaglutide (NNC0113-0217) in subjects with mild, moderate and severe degrees of hepatic impairment compared to subjects with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

* Subject with normal hepatic function or hepatic impairment (mild, moderate or severe)
* Body mass index (BMI) 18.5-40.0 kg/m^2 (both inclusive)

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using adequate contraceptive methods
* History of Crohn's disease, ulcerative colitis, or other inflammatory bowel disease
* Uncontrolled hypertension (defined as systolic blood pressure above or equal to 180 mmHg and/or diastolic blood pressure above or equal to 100 mmHg)
* Any donation of blood or plasma in excess of 400 mL within the 3 months preceding screening
* History of significant drug abuse, or a positive drug test at the screening visit (Visit 2)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-12-12 (Actual); Primary Completion 2015-01-12 (Actual); Study Completion 2015-01-12 (Actual)

PRIMARY OUTCOMES:
Area under the semaglutide plasma concentration curve | From time 0 to 24 hours after the 10th dosing

SECONDARY OUTCOMES:
Maximum observed semaglutide plasma concentration | 0 to 24 hours after the 10th dosing
Area under the SNAC (Sodium N-[8-(2-hydroxybenzoyl) amino] caprylate /salcaprozate sodium) plasma concentration time curve | From time 0 to 24 hours after the 10th dosing
Maximum observed SNAC plasma concentration | 0 to 24 hours after the 10th dosing

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (5):
- Novo Nordisk Investigational Site, Prague, Czechia
- Poland (3):
  - Novo Nordisk Investigational Site, Bialystok
  - Novo Nordisk Investigational Site, Warsaw
  - Novo Nordisk Investigational Site, Wołomin
- Novo Nordisk Investigational Site, Bratislava, Slovakia

REFERENCES:
- [Result] Baekdal TA, Thomsen M, Kupcova V, Hansen CW, Anderson TW. Pharmacokinetics, Safety, and Tolerability of Oral Semaglutide in Subjects With Hepatic Impairment. J Clin Pharmacol. 2018 Oct;58(10):1314-1323. doi: 10.1002/jcph.1131. Epub 2018 Apr 25. PMID 29693715
- [Derived] Overgaard RV, Navarria A, Ingwersen SH, Baekdal TA, Kildemoes RJ. Clinical Pharmacokinetics of Oral Semaglutide: Analyses of Data from Clinical Pharmacology Trials. Clin Pharmacokinet. 2021 Oct;60(10):1335-1348. doi: 10.1007/s40262-021-01025-x. Epub 2021 May 10. PMID 33969456
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com